CLINICAL TRIAL: NCT03271476
Title: EMDR Psychotherapy of Anxious-depressive Symptoms for Women That Present an Invasive Beast Cancer : a Faisability Study
Brief Title: EMDR Psychotherapy to Treat Anxious-depressive Symptoms in Breast Cancer Patient
Acronym: PSYCANCER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Collaborators: University of Lorraine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2017-01-CHRMT
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer; Eye Movement Desensitization and Processing; Psychoterapy
Keywords: Breast Cancer; EMDR
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: All the women will receive the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arms (Experimental): Experimental: EMDR psychotherapy All the women will be in this arm and thus will receive the same intervention which is : 8 sessions (1 per week). The first session is an inclusion visit at Metz-Thionville Hospital, then 6 EMDR psychotherapy sessions and finally a last visit one month after for data recovery (questionnaire and semi-directive interview)
  Interventions: Behavioral: EMDR psychotherapy

INTERVENTIONS:
Behavioral: EMDR psychotherapy — Visit 0 : patient inclusion (questionnaires and interview) Visit 1 : anamnesis Visit 2 : patient supporting Visit 3 : EMDR psychotherapy care Visit 4 : EMDR psychotherapy care Visit 5 : EMDR psychotherapy care and questionnaires Visit 6 : EMDR psychotherapy care Visit 7 : EMDR psychotherapy care Visit 8 : EMDR psychotherapy care ans questionnaires Visit 9 (one month after) : semi-directive interview and data recovery (questionnaires)

SUMMARY:
The study will consist in an adjustment/adaptation of the "standard EMDR protocol" for cancer disease, and most particulary for women who present a breast cancer and during adjuvant therapy. It will also test the faisability of the research, with a view to adjust the calendar and the ressources to put at disposal for a randomized control trial that follow. This study will also allow to test the need and acceptibility of this new psychotherapy for the patient, and to identify facilitators and obstacles : participation/rejection ratio, inclusion rythm, adhesion of the medical staff about the project

ELIGIBILITY:
Inclusion Criteria:

* Being a woman aged of 18 years or more
* Having a primary invasive breast cancer
* Having undergo a mastectomy for a primary invasive breast cancer
* Being able to complete the questionnaires
* Being informed of the study and having signed the informed consent
* Being affiliated to a welfare system

Exclusion Criteria:

* having contraindications to recieve EMDR psychotherapy (neurologic disorders, dissociatif states, oculomotor issues)
* Having started adjuvant treatments following surgery
* Having metastatic breast cancer
* Presenting physical polypathologies
* Having psychiatric antecedents (included anxiety and depressif disorders - assessed with M.I.N.I. (Sheehan and al., 1997)).
* Having drug or alcohol addiction
* Being placed under the safeguard of justice, guardianship or trusteeship
* Being pregnant or breast-feeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2018-07-25 (Actual)

PRIMARY OUTCOMES:
patients involvement | week 12
  acceptability of the new psychotherapy

SECONDARY OUTCOMES:
adequacy of the intervention with the field | Week 12
  adaptability of the EMDR protocol
EMDR psychotherapy efficacy during the study, we will survey our population several times with differents questionnaires | Week 12
  ratio of patients which wants to participate and effectively participate

CONTACTS AND LOCATIONS:
Overall Officials: Rafaele Longo, Dr, Principal Investigator — CHR Metz-Thionville
Locations (1):
- CHR Metz-Thionville, Metz, France

IPD SHARING:
Plan to Share IPD: Undecided